CLINICAL TRIAL: NCT07003451
Title: Novel Biomarkers in Assessment of Interstitial Lung Disease Associated With Rheumatoid Arthritis Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Waleed Gamal Elddin Khaleel, Assistant professor of chest diseases, Assiut University
Other Study IDs: RA-ILD-Associated-Biomarkers
Record Dates: First submitted 2025-05-26; First posted 2025-06-04 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Rheumatoid Arthritis; Interstitial Lung Disease
MeSH Terms: conditions — Arthritis, Rheumatoid; Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rheumatoid Arthritis with ILD: Rheumatoid arthritis patients with interstitial lung disease diagnosed by high resolution CT and correlated to level of biomarkers
  Interventions: Diagnostic Test: Calprotectin Level

INTERVENTIONS:
Diagnostic Test: Calprotectin Level — Measurement of calprotectin level to presence and severity of ILD asessed via Warrick's score

SUMMARY:
- Assess Krebs von den Lungen-6 (KL-6) and Calprotectin as novel biomarkers for diagnosis of ILD among Rheumatoid arthritis patients

DETAILED DESCRIPTION:
Rheumatoid arthritis (RA) is a systemic autoimmune disease characterized by small joint synovitis that is estimated to affect 0.3% to 1% of the global population. Extraarticular disease may occur in up to 50% of patients with RA, with pulmonary manifestations among the most common extraarticular features. Interstitial lung disease (ILD) clinically affects up to 10% of patients with RA and subclinically affects up to 40%.

RA-ILD typically presents as a usual interstitial pneumonia (UIP) or nonspecific interstitial pneumonia pattern. Diagnosis requires a thorough evaluation, including laboratory and imaging studies; pulmonary function testing (PFT); medication review; occasionally, tissue histopathology; and frequently, multidisciplinary input.

Prompt recognition of RA-ILD is crucial because it warrants close monitoring and often necessitates therapeutic alterations.

Biomarkers are a promising area of investigation in RA-ILD because they have the potential to advance pathophysiologic understanding and elucidate therapeutic targets, improve disease identification and diagnostic accuracy, facilitate prognostication, and inform treatment decisions. Although imaging and histopathology have important roles that are unlikely to be replaced by biomarkers, they can be nonspecific in RA-ILD, can be impractical to obtain in certain settings, and cannot be scaled for population health efforts.

Calprotectin belongs to the S-100 proteins produced by neutrophils, which likely contribute to idiopathic pulmonary fibrosis (IPF) pathogenesis. Calprotectin is a well-established biomarker in inflammatory bowel diseases.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Rheumatoid arthritis, age > 18 years.

Exclusion Criteria:

* Patients who refuse to participate in the study,
* Patients with evidence of worsening or exacerbation of RA over the previous 6 months,
* concomitant diagnosis of an active neoplasia, or
* patients who had previously received radiotherapy,
* End organ failure.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Confirmed diagnosis of Rheumatoid arthritis, age > 18 years and confirmed diagnosis of ILD based on HRCT findings and Pulmonary function test results.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
calprotectin level among rheumatoid arthritis patients with interstitial lung disease | day 1
  calprotectin level among rheumatoid arthritis patients with interstitial lung disease

CONTACTS AND LOCATIONS:
Overall Officials: waleed gamal elddin, ass. prof, Principal Investigator — Assiut University
Locations (1):
- Assiut University hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Furukawa H, Oka S, Higuchi T, Shimada K, Hashimoto A, Matsui T, Tohma S. Biomarkers for interstitial lung disease and acute-onset diffuse interstitial lung disease in rheumatoid arthritis. Ther Adv Musculoskelet Dis. 2021 Jun 18;13:1759720X211022506. doi: 10.1177/1759720X211022506. eCollection 2021. PMID 34211592
- [Background] Machahua C, Guler SA, Horn MP, Planas-Cerezales L, Montes-Worboys A, Geiser TK, Molina-Molina M, Funke-Chambour M. Serum calprotectin as new biomarker for disease severity in idiopathic pulmonary fibrosis: a cross-sectional study in two independent cohorts. BMJ Open Respir Res. 2021 Jan;8(1):e000827. doi: 10.1136/bmjresp-2020-000827. PMID 33451989